CLINICAL TRIAL: NCT02584192
Title: Efficacy of Early Home-based Cardiac Rehabilitation Program for Patients After Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lin Xu (Other)
Responsible Party: Sponsor-Investigator, Lin Xu, M.D., Guangzhou General Hospital of Guangzhou Military Command
Organization: Guangzhou General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR2014
Record Dates: First submitted 2015-10-16; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the rehabilitation group (Experimental): entailing an early home-based CR program
  Interventions: Behavioral: entailing an early home-based CR program
- the control group (Other): enter the usual care program, including the importance of carrying out physical activity, which was performed during inpatient care.
  Interventions: Other: enter the usual care program

INTERVENTIONS:
Behavioral: entailing an early home-based CR program — enter the early outpatient phase of CR program. The progressive exercise training of this phase was performed without supervision after their discharge. The CR program consisted of a five-minute warm-up period (stretching), a twenty-minute aerobic exercise (walking or trotting, gymnastics), and a five-minute cooling-down period (stretching)
  Arms: the rehabilitation group
Other: enter the usual care program — enter the usual care program, including the importance of carrying out physical activity, which was performed during inpatient care.
  Arms: the control group

SUMMARY:
The purpose of this study was to evaluate the effect of this CR program on the improvement of myocardial function using the three-dimensional speckle tracking echocardiography (3D-STE) in AMI patients.

DETAILED DESCRIPTION:
The effect of early short-term home-based cardiac rehabilitation (CR) program on left ventricular function in acute myocardial infarction (AMI) patients is not clear yet.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18-65 years with a confirmed AMI diagnosis
* Being suitable for the CR program
* Undergoing PCI at the entry

Exclusion Criteria:

* Known ischemic heart disease, heart valvular lesions, intra-ventricular conduction disturbances, malignant arrhythmia, cardiac shock, and poor echocardiographic conditions to take STE examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
myocardial function using the three-dimensional speckle tracking echocardiography (3D-STE) | Change from baseline strain parameters at four-week follow-up

REFERENCES:
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536